CLINICAL TRIAL: NCT06791512
Title: mFOLFOX6 + Bevacizumab + PD-1 Monoclonal Antibody Versus mFOLFOX6 as Neoadjuvant Therapy for Locally Advanced pMMR/MSS Colorectal Cancer: A Prospective, Multicenter, Randomized Phase III Study (BASKETIII)
Brief Title: mFOLFOX6 + Bevacizumab + PD-1 Monoclonal Antibody Vs. mFOLFOX6 in Locally Advanced pMMR/MSS CRC
Acronym: BASKETⅢ
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jun Huang (Other)
Responsible Party: Sponsor-Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2024365
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer (CRC); pMMR/MSS Adenocarcinoma of the Colon or Rectum
Keywords: Colorectal cancer; pMMR/MSS; Neoadjuvant Therapy; PD-1 monoclonal antibody; mFOLFOX6
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant therapy of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody (Experimental): Participants will receive the first five doses of neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and a 48-hour continuous infusion of 5-fluorouracil 2400 mg/m2) combined with sintilimab (200 mg, intravenous) and Bevacizumab (5 mg/kg, intravenous). The sixth dose will consist of the same regimen of mFOLFOX6 and PD-1 monoclonal antibody, but not plus bevacizumab, in order to allow sufficient withdrawal time of Bevacizumab for surgery.
  Interventions: Drug: mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody
- Neoadjuvant therapy of mFOLFOX6 (Active Comparator): Participants will receive the neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and a 48-hour continuous infusion of 5-fluorouracil 2400 mg/m2).
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody — Participants in the experimental group will receive the neoadjuvant therapy regimen of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody. And the first five doses received the neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and 5-fluorouracil 2400 mg/m2 continuous pumping for 48 hours) combined with sintilimab (200 mg, intravenous) and Bevacizumab (5 mg/kg, intravenous), and the sixth dose received the same regimen of mFOLFOX6 and PD-1 monoclonal antibody but not plus bevacizumab, in order to allow sufficient withdrawal time of Bevacizumab for surgery.
  Other Names: mFOLFOX6
  Arms: Neoadjuvant therapy of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody
Drug: mFOLFOX6 — Participants in the control group will receive the neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and 5-fluorouracil 2400 mg/m2 continuous pumping for 48 hours) alone.
  Other Names: mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody
  Arms: Neoadjuvant therapy of mFOLFOX6

SUMMARY:
Neoadjuvant immunotherapy has shown promising therapeutic effects in mismatch repair-deficient or microsatellite instability-high (dMMR/MSI-H) colorectal cancer (CRC). However, for patients with mismatch repair-proficient or microsatellite stable (pMMR/MSS) CRC, the efficacy of PD-1 monoclonal antibody remains limited. Enhancing the efficacy of immunotherapy in pMMR/MSS CRC has become a key area of exploration. Additionally, for locally advanced (cT4NxM0) CRC patients, achieving R0 resection poses a significant challenge. Failure to achieve R0 resection often results in recurrence, severely impacting patient survival outcomes. Our previous phase II clinical study (BASKET Ⅱ) demonstrated that the neoadjuvant regimen of mFOLFOX6 combined with Bevacizumab and PD-1 monoclonal antibody significantly enhanced the immunotherapy sensitivity of locally advanced pMMR/MSS CRC, leading to improved pathological complete response (pCR) rates and higher R0 resection rates. This prospective, multicenter, randomized phase III trial aims to evaluate whether the neoadjuvant regimen of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody can further improve pCR rate, enhance survival outcomes, and maintain an acceptable safety profile compared to mFOLFOX6 alone in pMMR/MSS locally advanced CRC patients.

DETAILED DESCRIPTION:
This clinical trial is an open-label, prospective, multicenter, randomized phase III study. The aims of this study are to evaluate whether the the neoadjuvant regimen of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody can improve the pathological complete response (pCR) rate, enhance survival outcomes, and maintain manageable toxicity compared to mFOLFOX6 alone in patients with locally advanced pMMR/MSS CRC. Eligible participants will be randomly assigned in a 1:1 ratio to either the experimental group or the control group. Participants in the experimental group will receive the neoadjuvant therapy regimen of mFOLFOX6 + Bevacizumab + PD-1 monoclonal antibody. And the first five doses will receive the neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and a 48-hour continuous infusion of 5-fluorouracil 2400 mg/m2) combined with sintilimab (200 mg, intravenous) and Bevacizumab (5 mg/kg, intravenous). The sixth dose will consist of the same regimen of mFOLFOX6 and PD-1 monoclonal antibody, but not plus bevacizumab, in order to allow sufficient withdrawal time of Bevacizumab for surgery. Participants in the control group will receive the neoadjuvant therapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and a 48-hour continuous infusion of 5-fluorouracil 2400 mg/m2) alone. Subjects in both the experimental and control groups will undergo radical surgical treatment after completing the neoadjuvant therapy. Those achieving pCR based on postoperative pathology will be regularly followed up according to the follow-up protocol. Participants who do not achieve pCR will receive six cycles of adjuvant therapy after surgery, followed by regular follow-up assessments as outlined in the protocol after completing the final cycle of adjuvant therapy. The primary outcome of this study is to evaluate the 3-year disease-free survival (DFS). Secondary objectives include the pCR rate, major pathological response (MPR) rate, neoadjuvant therapy-related toxicities, R0 resection rate, tumor downstaging rate, and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the colon or upper rectum.
2. Tumor biopsy immunohistochemical (IHC) identified pMMR, including all of the MSH1,MSH2,MSH6 and PMS2 protein expression and diagnosed as proficient mismatch repair(pMMR), or microsatellite stable (MSS) identified through next-generation sequencing or polymerase chain reaction.
3. Clinical staging of cT4NxM0, with or without positive mesorectal fascia (MRF), and with or without extramural vascular invasion (EMVI); imaging confirms that the lower margin of the tumor is located above the peritoneal reflection (colon or upper rectum).
4. Staging method: All patients must undergo chest, abdominal, and pelvic contrast-enhanced CT, rectal palpation, and high-resolution MRI. Positive perienteric lymph nodes (LNs) are defined as LNs with a short diameter ≥10 mm or LNs exhibiting typical metastatic shape and MRI characteristics. When staging results are contradictory, clinical data must be re-evaluated and confirmed by the central evaluation group. Distant metastases must be excluded through chest and abdominal contrast-enhanced CT and pelvic contrast-enhanced MRI.
5. No symptoms of intestinal obstruction, or obstruction successfully relieved by proximal colostomy.
6. No history of colorectal surgery.
7. No prior chemotherapy or radiotherapy.
8. No history of biopharmaceutical treatments (e.g., monoclonal antibody ), immunotherapy (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies), or treatment with investigational drugs.
9. Endocrine therapy history: Not restricted.
10. Signed informed consent obtained.

Exclusion Criteria:

1. Arrhythmias requiring anti-arrhythmic treatment (except β-blockers or Digoxin), symptomatic coronary artery disease, myocardial ischemia (myocardial infarction within the past 6 months), or congestive heart failure (CHF) > NYHA Class II.
2. Severe hypertension that is not well controlled by medication.
3. History of HIV infection or active chronic Hepatitis B or C (with high viral DNA load).
4. Active tuberculosis (TB), ongoing anti-TB treatment, or anti-TB treatment within 1 year prior to trial screening.
5. Other active severe infections as defined by NCI-CTCAE v5.0.
6. Evidence of distant metastasis beyond the pelvic region.
7. Blood dyscrasias or organ dysfunction.
8. History of pelvic or abdominal radiotherapy.
9. Multiple colorectal cancer or multiple primary tumors.
10. Epilepsy requiring treatment (e.g., steroids or anti-epileptic drugs).
11. History of other malignancies within the past 5 years.
12. History of drug abuse, or medical, psychological, or social conditions that could interfere with patient participation or the evaluation of study results.
13. Any active autoimmune disease or a history of autoimmune disease (including but not limited to interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators).
14. Administration of any live attenuated vaccine within 4 weeks prior to inclusion.
15. Long-term use of immunosuppressants or systemic/topical corticosteroids (dose >10 mg/day prednisolone or equivalent).
16. Known or suspected allergy to any study-related drug.
17. Any unstable condition that could compromise patient safety or compliance.
18. Pregnant or breastfeeding women, or women of childbearing potential not using effective contraception.
19. Refusal to provide signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
3 years DFS Rate | 3 years
  3 years Disease Free Survival Rate

SECONDARY OUTCOMES:
pCR rate | 1 year
  pathological complete response rate
MPR rate | 1 year
  major pathologic response
Toxicities Associated with Neoadjuvant Therapy | 1 year
  Incidence of adverse events related to neoadjuvant therapy as assessed by CTCAE v5.0
R0 resection rate | 1 year
  R0 resection rate in participants
Down-stage rate | 1 year
  Down-stage rate of pathological stage after surgery compared with clinical stage before neoadjuvant therapy
3 years OS Rate | 3 years
  3 years Overall Survival Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No